CLINICAL TRIAL: NCT03591757
Title: An Open-Label, Investigator Study to Evaluate the Short-term (4 Weeks) Effects of TOLCAPONE on Transthyretin Stability in Subjects With Leptomeningeal TTR Amyloidosis (ATTR) With and Without CNS Manifestations
Brief Title: Short-term Effects of TOLCAPONE on Transthyretin Stability in Subjects With Leptomeningeal TTR Amyloidosis (ATTR)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Corino Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, John L. Berk, Associate Professor,Dept of Medicine, Amyloidosis Center, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-37757
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Transthyretin Amyloidosis; Amyloidosis, Leptomeningeal, Transthyretin-Related
Keywords: Tolcapone; Transthyretin (TTR); Mutant TTR; Plasma TTR; CSF TTR; Tetramer stability; Leptomeningeal; Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis | interventions — Tolcapone

STUDY DESIGN:
Intervention Model Description: Patients with hATTR mutations conferring leptomeningeal amyloidosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tolcapone (Experimental): Tolcapone will be administered to assess the short-term (4 weeks) effects on plasma and CSF TTR tetramer stability in subjects with TTR CNS Amyloidosis. Tolcapone is currently licensed for the treatment of Parkinson's disease in combination with levodopa/carbidopa. It is an immediate release product and is currently used at either 100 mg or 200 mg three times a day during waking hours. During this trial, participants will be taking 100mg for 14 days, and then 200mg for 14 days.
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Drug: Tolcapone — Tolcapone will be administered at 300 mg/day (100mg TID) orally to participants for 14 days and then 600 mg/day (200 mg TID) orally to participants for 14 days (approximately 5 hours apart). Participants will initiate 200mg TID after blood collection on Day 14.
  Other Names: Tasmar

SUMMARY:
The purpose of this study is to determine whether Tolcapone crosses from the blood stream into the fluid around the brain and stabilizes the protein that makes leptomeningeal amyloid. Tolcapone is a commercially available generic drug that treats Parkinson's disease.

The Investigator plans to evaluate Tolcapone as a treatment for ATTR (Transthyretin Amyloidosis), a rare genetic disease often causing death within 5-15 years after diagnosis. ATTR is characterized by deposition of misfolded protein known as amyloid, in one or more organ systems (including the peripheral and autonomic nervous systems, the heart, the brain and the eyes). The age at which symptoms begin to develop varies widely ranging between 20 to 70 years old. ATTR is progressive, and some variants can have a fatal outcome within a few years of presentation. Treatment options include supportive and symptomatic care that may slow or stop progressive decline in functional state but do not alter the pathological process. Liver transplant can be performed in selected patients but is limited by organ supply, requires lifelong immunosuppression, and may be complicated by progressive heart and nerve amyloid deposition. Importantly, liver transplant does not alter the natural course of central nervous system amyloid disease. To date, no treatment for ATTR penetrates the CNS.

At present there is no FDA approved treatment for ATTR amyloidosis in the US. In Europe, Tafamidis has been approved for treatment of stage 1 ATTR-polyneuropathy since 2012. Tafamidis and Tolcapone bind to the thyroxine binding site of TTR (with different drug-transthyretin interactions) and in so doing stabilizes the tetrameric form of TTR, preventing dissociation and amyloid fibril formation The preclinical and clinical data from a variety of experimental systems support the therapeutic activity of TOLCAPONE in TTR mediated disease.

DETAILED DESCRIPTION:
This study is designed as a clinical proof-of-concept evaluating whether TOLCAPONE is capable of stabilizing tetrameric TTR (Transthyretin) in the plasma and CSF of symptomatic or asymptomatic patients with leptomeningeal ATTR. Additionally the study will determine the plasma and CSF concentrations of TOLCAPONE needed to induce maximal stabilization of TTR across different TTR variants (TTR mutations).

The study will be carried out in two different populations of subjects, defined by the TTR variant expressed:

* Mutant TTR (up to 10 subjects): symptomatic leptomeningeal TTR patient with any documented leptomeningeal mutations in the TTR gene.
* Mutant TTR (remaining subjects up to 10): asymptomatic leptomeningeal TTR patient with any documented leptomeningeal mutation in the TTR gene.

TTR tetramers stability in plasma and CSF samples will be determined by urea-induced denaturation methodology.

ELIGIBILITY:
Inclusion Criteria:

* Genotyping of variant TTR
* Documented CNS manifestation or expression of variant TTR with leptomeningeal potential

Exclusion Criteria:

* Patients who are unable to provide informed consent
* Contraindication for Tolcapone
* An ALT or AST measurement > 2 times the ULN (Upper Limit of Normal)
* Estimated glomerular filtration rate (eGFR) ≤ 25 ml/min/1.72M2
* Treatment with a known TTR tetramer protein stabilizer within the last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Change in plasma TTR stabilization | pre-treatment (Day 0) and Day 28
  TTR stabilization will be measured in plasma samples from each participant before the first dose of study drug and 2 hours after the last 100 mg study drug dose.
Change in CSF TTR stabilization | pre-treatment (Day 0) and Day 28
  TTR stabilization will be measured in CSF samples obtained from each participant before the first dose of study drug and 2 hours after the last 200 mg dose.

SECONDARY OUTCOMES:
Changes in plasma TTR stabilization | pre-treatment (Day 0) and Day 14
  TTR stabilization will be measured in plasma samples from each participant before the first dose of study drug and 2 hours after the day 14 study drug dose.
Changes in plasma TTR stabilization | Day 14 and Day 28
  TTR stabilization will be measured in plasma samples from each participant 2 hours after the day 14 study drug dose.and 2 hours after the 28 day study dose
Tolcapone Concentration in CSF | Day 14
  Tolcapone concentration will be measured in CSF at Day 14 prior to starting 200mg TID dosing.
Tolcapone Concentration in CSF | Day 28
  Tolcapone concentration will be measured in CSF at Day 28 2 hours after dose
Tolcapone Concentration in Serum | Day 14
  Tolcapone concentration will be measured in serum at Day 14 prior to initiating 200 mg TID dosing
Tolcapone Concentration in Serum | Day 28
  Tolcapone concentration will be measured in serum at Day 28 2 hours after last dose

CONTACTS AND LOCATIONS:
Overall Officials: John L Berk, MD, Principal Investigator — The Amyloidosis Center, BUSM
Locations (1):
- Amyloidosis Center, Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No